CLINICAL TRIAL: NCT04091828
Title: Assessment of Cognitive Functions in Bipolar Disorder Patients
Brief Title: Assessment of Cognitive Functions in Bipolar Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Salama Ahmed Omar, Assessment of cognitive function in bipolar patients, Assiut University
Other Study IDs: cognition in bipolar patients
Record Dates: First submitted 2019-09-05; First posted 2019-09-17 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biplar patients: diagnosed by DSM-5 and divided to manic,depressed and mixed last episod
- controlled subject: not have any medical or psychatric problem affect cognition

SUMMARY:
Assessment of cognitive function in manic bipolar patient

DETAILED DESCRIPTION:
Assessment of severity of mania and depression in bipolar patients then evaluate their cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Of both sex
* Diagnosed as bipolar by DSM-5(patient)

Exclusion Criteria:

* Current medical and psychiatric comorbidities which may affect cognitive status.
* Substance abuse or dependence (except nicotine and caffeine)in last month.
* Somatic treatment with drugs known to affect cognitive status (cortisol, antihistamines, etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: stable people not irritable
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of severity of mania in bbipolar patients | 2019-2022
  EVALUATE manic patients by Young Mania Rating Scale (YMRS)
Assessment of severity of depression in bipoiar patients | 2019-2022
  Evaluate depressed patients by Hamilton Rating Scale for depression(HRS).
Assessment of cognitive function in bipoiar patients | 2019-2022
  Evaluate cognition in included patients by Montreal Cognitive Assessment(MOCA) and P300.

SECONDARY OUTCOMES:
Correlation between cognitive state in bipolar patient and(onset age,illness duration and number of episodes). | 2019-2021
  from history